CLINICAL TRIAL: NCT02712736
Title: Quality of Life in Primary Sclerosing Cholangitis
Brief Title: Quality of Life in Patients With Primary Sclerosing Cholangitis
Acronym: QOL in PSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00069683
Record Dates: First submitted 2016-03-11; First posted 2016-03-18 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey respondents (Other): The patients who consent to participate will be sent home from the clinic with a survey to complete and return via mail in a provided addressed, stamped envelope. The survey consists of the Short Form-36 (SF-36), the Chronic Liver Disease Questionnaire (CLDQ), questions from the PROMIS SexFs v2.0, questions regarding perceived risk for liver transplant, cholangiocarcinoma, and colorectal carcinoma, as well as perceived overall life expectancy, and questions regarding complementary and alternative medicine use.
  Interventions: Other: quality of life survey

INTERVENTIONS:
Other: quality of life survey — subjects with PSC will be administered a survey to assess their quality of life

SUMMARY:
The purpose of this study is to assess the healthcare-related quality of life (HRQOL), the impact of risk of liver transplant and risk of malignancy on HRQOL, and the complementary and alternative medicine use in patients with PSC.

DETAILED DESCRIPTION:
A cohort of adult (age ≥ 18) patients with a diagnosis of PSC will be identified. The patients will be approached about participating in the study while at their appointment, either by the investigators or someone else known to the patient. If the patient agrees, the investigators or other key personnel will then provide information about the study and obtain their informed consent to participate.

The patients who consent to participate will be sent home from the clinic with a survey to complete and return via mail in a provided addressed, stamped envelope. The survey consists of the Short Form-36 (SF-36), the Chronic Liver Disease Questionnaire (CLDQ), questions from the PROMIS SexFs v2.0, questions regarding perceived risk for liver transplant, cholangiocarcinoma, and colorectal carcinoma, as well as perceived overall life expectancy, and questions regarding complementary and alternative medicine use.

Demographic information and clinical data will also be obtained from the patient's electronic medical record. The study will be cross-sectional in nature, and there will be no follow-up with the subjects after the survey is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18) patients with PSC, confirmed by laboratory tests, imaging, and/or liver biopsy

Exclusion Criteria:

* Patients <18
* Patients who have undergone liver transplant, patients with frank hepatic encephalopathy
* Patients with active inflammatory bowel disease (IBD) flares
* Patients with malignancies
* Patients unable to understand English
* Patients refusing to participate or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-09-22 (Actual)

PRIMARY OUTCOMES:
Impaired quality of life as measured by questionnaire | Approximately 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Muir, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No